CLINICAL TRIAL: NCT01662765
Title: Conservative Versus Surgical Treatment of Umbilical Pilonidal Sinus Disease: A Prospective, Randomised, and Multicenter Clinical Trial
Brief Title: Conservative Versus Surgical Treatment of Umbilical Pilonidal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Park Gaziantep Hospital (Other)
Collaborators: Zeugma Saglik Hizmetleri San. Tic. Ltd. Sti. (Industry)
Responsible Party: Principal Investigator, Mehmet Kaplan, Principal investigator, Medical Park Gaziantep Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MK-003-UPS
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2016-12

CONDITIONS: Pilonidal Sinus; Sinus; Dermal, Pilonidal; Umbilical Granuloma
Keywords: Umbilical pilonidal sinus; Treatment; Surgery; Conservative; Investigational treatment; After care
MeSH Terms: conditions — Pilonidal Sinus; Fistula | interventions — Surgical Procedures, Operative; Conservative Treatment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery (Experimental): Circular incision 2-3 mm below the skin level in the umbilicus through the subcutaneous fat towards the linea alba. Dissection of the subcutaneous tissue within the umbilicus and its deep connection to preperitoneal fat through the linea alba. Excision of the umbilical complex containing pilonidal cyst 3 mm below the umbilical ostium.
  Approximation of the subcutaneous tissue with a single purse-string absorbable suture. The specimen, including the umbilical complex (pilonidal cyst, and involved skin and subcutaneous tissue), was transferred to department of pathology for histopathological examination.
  Interventions: Procedure: Surgery
- Conservative (Active Comparator): Conservative treatment described as follow:
  Under local anesthesia, extracting all protruding hair, and curetting the granulation tissue and pilonidal cyst deep in the umbilicus.
  postoperative management include antibiotic treatment with ampicilline plus sulbactam and ornidazole, shaving surrounding skin, washing twice daily, and keeping umbilicus dry.
  Interventions: Other: conservative

INTERVENTIONS:
Procedure: Surgery — modified umbilectomy
  Other Names: umbilectomy
  Arms: Surgery
Other: conservative — this treatment will include conservative procedures under local anesthesia for patient comfort.
  Other Names: non-surgical management
  Arms: Conservative

SUMMARY:
The aim of the study was to compare the results of conservative and surgical treatment, to create an algorithm for the management of the disease, and gain more information about the etiology, pathogenesis, and course of the disease. The investigators hypothesise that surgical treatment of UPS will be better than conservative management in terms of recurrence rate, healing time, patient comfort and satisfaction, and cost effectiveness.

DETAILED DESCRIPTION:
Because of its rarity, umbilical pilonidal sinus (UPS) is still poorly understood in terms of diagnosis, etiology, and the best treatment options.

UPS is thought caused by hair penetrating the skin, leading to a foreign-body reaction and development of a sinus lined with granulation tissue. Most of the patients complain of pain, discharge or bleeding from the umbilicus when symptoms develop. It can be diagnosed with a careful examination, in which hairs can be seen deep in the umbilicus and usually protrude from a small sinus.

Regarding the optimal treatment of the disease, a complete consensus has not yet been achieved. Some publications are recommended conservative treatment, while surgical treatment is recommended in others.

A more meaningful comparison of the two modalities is that of a randomized controlled trial. We, therefore, present our data of prospective randomized controlled clinical trial comparing conservative versus surgical treatment of UPS.

This was a multicenter, prospective balanced randomization, double blind, active-controlled, parallel-group, superiority study conducted in Turkey, under the direction of a principal investigator (MK). Eligible patients with UPS were randomized for either conservative treatment (CT) or surgical treatment (ST), and then the results of both groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* all patients willing to participate to the study with the diagnosis of umbilical pilonidal sinus

Exclusion Criteria:

* no informed consent
* serious coagulation abnormalities
* known allergy to local anesthetics
* pregnancy, or women who refused contraception at the time of treatment
* other concomitant umbilical pathologies such as umbilical hernia, granuloma, dermoid cyst
* the patients who diagnosed with urachal and omphalomesenteric anomalies through radiological investigation
* patients who underwent umbilical operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2003-11; Primary Completion 2010-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet KAPLAN, MD, Principal Investigator — Medical Park Gaziantep Hospital, Gaziantep, Turkey
Locations (5):
- Turkey (Türkiye) (5):
  - Hatem Hospital, Gaziantep
  - Medical Park Gaziantep Hospital, Gaziantep
  - 25 Aralık Familiy Physician Health Center, Gaziantep
  - Dr.Ersin Arslan State Hospital, Gaziantep
  - Şehitkamil State Hospital, Gaziantep

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaplan M, Ozcan O, Kaplan FC, Yalcin HC, Salman B. Conservative vs Surgical Interventions for Umbilical Pilonidal Sinus: A Multicenter, Double-Blind, Prospective, Randomized Clinical Trial. J Am Coll Surg. 2016 May;222(5):878-89. doi: 10.1016/j.jamcollsurg.2016.01.056. Epub 2016 Feb 23. PMID 27016906

RESULTS

PARTICIPANT FLOW:
Groups:
- Conservative: Conservative treatment described as follow:
  Under local anesthesia, extracting all protruding hair, and curetting the granulation tissue and pilonidal cyst deep in the umbilicus.
  postoperative management include antibiotic treatment with ampicilline plus sulbactam and ornidazole, shaving surrounding skin, washing twice daily, and keeping umbilicus dry.
  conservative: this treatment will include conservative procedures under local anesthesia for patient comfort.
Period: Overall Study
Arm/Group | Conservative | Surgery
Started | 42 | 42
Completed | 41 | 40
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conservative | Surgery | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 21.80 [12 to 34] | 19.86 [10 to 37] | 20.83 [10 to 37]
Gender [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 39 | 40 | 79
Region of Enrollment [Number; unit: participants]
  Turkey | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate
Description: Primary outcome was the cure rate. Absence of recurrence within two year after the first treatment was considered as a cure.
  Recurrence was defined as the appearance of a new, active discharging sinus or granulation tissue with/without a bit of hairs in the deep of the umbilicus within two years after therapy.
Time Frame: 2 year after initial treatment
Population: Of the 84 patients 41 patients in the CT group. and 40 patients in ST group were analyzed
Measure: Number; unit: participants
Arm/Group | Conservative | Surgery
Number analyzed (Participants) | 41 | 40
participants | 28 | 40

2. Secondary Outcome: Healing Time
Description: the time form initial treatment to healing the wound and/or sinus and/or granulation tissue and no any sign of drainage with no longer need for dressing and wound care in either treatment arms.
Time Frame: two year
Measure: Mean (Standard Deviation); unit: days
Groups:
- Surgery: Circular incision 2-3 mm below the skin level in the umbilicus through the subcutaneous fat towards the linea alba. Dissection of the subcutaneous tissue within the umbilicus and its deep connection to preperitoneal fat through the linea alba. Excision of the umbilical complex containing pilonidal cyst 3 mm below the umbilical ostium.
  Approximation of the subcutaneous tissue with a single purse-string absorbable suture. The specimen, including the umbilical complex (pilonidal cyst, and involved skin and subcutaneous tissue), was transferred to department of pathology for histopathological examination.
  Surgery: modified umbilectomy
Arm/Group | Surgery | Conservative
Number analyzed (Participants) | 42 | 42
days | 12.81 (2.96) | 17.06 (5.1)

3. Secondary Outcome: Visual Analogue Scale for Patient Satisfaction (VAS-PS)
Description: Well-being and satisfaction scales comprised linear metric scales known as "visual analogue scales," with grades from 0 (worst imaginable health state and extremely dissatisfied with the treatment) to 100 (best imaginable health state and extremely satisfied with the treatment).
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Conservative: Conservative treatment described as follow:
  Under local anesthesia, extracting all protruding hair, and curetting the granulation tissue and pilonidal cyst deep in the umbilicus.
- Surgery: Circular incision 2-3 mm below the skin level in the umbilicus through the subcutaneous fat towards the linea alba. Dissection of the subcutaneous tissue within the umbilicus and its deep connection to preperitoneal fat through the linea alba. Excision of the umbilical complex containing pilonidal cyst 3 mm below the umbilical ostium.
Arm/Group | Conservative | Surgery
Number analyzed (Participants) | 33 | 42
units on a scale | 66 (8) | 71 (6)

4. Other Pre Specified Outcome: Costs
Description: from initial treatment to the complete healing, all kind of cost will be calculated.
Time Frame: two year
Measure: Mean (Standard Deviation); unit: USD dollars
Groups:
- Surgery: Excision of the umbilical complex containing pilonidal cyst 3 mm below the umbilical ostium.
Arm/Group | Conservative | Surgery
Number analyzed (Participants) | 42 | 42
USD dollars | 609 (224) | 479 (75)

ADVERSE EVENTS:
Groups:
- Surgery: Circular incision 2-3 mm below the skin level in the umbilicus through the subcutaneous fat towards the linea alba. Dissection of the subcutaneous tissue within the umbilicus and its deep connection to preperitoneal fat through the linea alba. Excision of the umbilical complex containing pilonidal cyst 3 mm below the umbilical ostium.
  Approximation of the subcutaneous tissue with a single purse-string absorbable suture.
Arm/Group | Conservative | Surgery
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No